CLINICAL TRIAL: NCT06217835
Title: Changes in Activity of Erector Spinae and Gluteus Medius Muscles With the Presence of Simulated Lower Limb Dysmetria
Brief Title: What Are the Effects of Lower Limb Dysmetria on Gluteus Medius and Erector Spinae Musculature?
Acronym: s-EMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CamiloJcU-Fisio
Record Dates: First submitted 2023-12-04; First posted 2024-01-23 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Muscular Disorders, Atrophic
Keywords: Low Back Pain; electromyography; Leg Length Inequality; lower limb length
MeSH Terms: conditions — Muscular Disorders, Atrophic; Low Back Pain; Leg Length Inequality

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0,5 cm jig (Experimental): A template with the dimensions indicated is introduced to the user and he/she walks for 1 minute.
  Interventions: Other: To evaluate the response of an orthopedic insole; Other: evaluate activation of musculature
- 1 cm jig (Experimental): A template with the dimensions indicated is introduced to the user and he/she walks for 1 minute.
  Interventions: Other: To evaluate the response of an orthopedic insole; Other: evaluate activation of musculature
- 1,5 cm jig (Experimental): A template with the dimensions indicated is introduced to the user and he/she walks for 1 minute.
  Interventions: Other: To evaluate the response of an orthopedic insole; Other: evaluate activation of musculature

INTERVENTIONS:
Other: To evaluate the response of an orthopedic insole — To evaluate the response of an orthopedic insole of different heights on gait.
Other: evaluate activation of musculature — To evaluate the response caused by an orthopedic insole of different heights on the indicated musculature.

SUMMARY:
Gluteus Medius (GM) has also been implicated in the development of Low Back Pain (LBP). GM is one of the main pelvic, where he actively participates in control of motion in the frontal and transverse plane, and hip , improving stability to the lumbopelvic-hip complex.

The aim of present study was to investigate whether modifying lower limb length with a different foot insoles of 0.5, 1 and 1.5 cm in a normal population has an effect on ES and GM activity and as a consequence in LBP. As a secondary objective, in turn, to evaluate whether ES and GM activity has an effect on jumping ability as assessed through CMJ.

DETAILED DESCRIPTION:
Background: Length leg discrepancy (LLD), regardless of its origin, is a very common pathology that can contribute to low back pain. Various authors point out its relationship with the lack of activation of both the gluteus medius (GM) and the ipsilateral erector spinae (ES). The purpose of this study was to identify the activation of Es and GM with different simulated LLD, correlating said activation with the LBP. In turn, to evaluate whether ES and GM activity has an effect on jumping ability as assessed through CMJ. (2) Method: a sample of healthy subjects was selected to whom an artificial LLD was incorporated through a 0.5, 1 and 1.5 cm insole, measuring with EMGs in these 3 moments while walking and performing a counter movement jump (CMJ). The measurement was carried out in random order, in terms of insole height, using a Latin Square. Muscle activation patterns were recorded for 30 seconds at each of the insole heights while walking at 5.7 km/h and compared with the maximum voluntary contraction (MVC), both on the ipsilateral and contra-lateral sides. These muscles were then measured under the same circumstances during the development of the CMJ. (3)

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* The volunteers had no problems in range of motion of joints of the lower limbs
* pelvic obliquity due to a functional leg length discrepancy.
* obesity with body mass index (BMI) 35 > kg/m²

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Height CMJ | 1 week
  CMJ jump flight height
Height DJ LEFT | 1 week
  Flying height in drop jump left leg
Height DJ RIGHT | 1 week
  Flying height in drop jump right leg
Gluteus medius (mv) | 1 week
  Gluteus medius activation (mv)
Erector Spinae (mv) | 1 week
  Erector Spinae activation (mv)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Cimadevilla, PT, Study Director — Camilo Jose Cela University
Locations (1):
- Juan Hernández Lougedo, Villanueva de la Cañada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No